CLINICAL TRIAL: NCT04080830
Title: Patient Registration Study of Acute Ischemic Stroke/Transient Ischemic Attack(TIA ) With Atrial Fibrillation
Brief Title: Registration Study of Acute Ischemic Stroke/Transient Ischemic Attack (TIA) With Atrial Fibrillation
Acronym: AISWAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Sufang Xue, principal investigator, Xuanwu Hospital, Beijing
Other Study IDs: ID-8849
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation
Keywords: Registration Study; Acute Ischemic Stroke; Atrial Fibrillation
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute ischemic stroke/transient ischemic attack (TIA) with AF: patients with Acute ischemic stroke/TIA and Atrial fibrillation (observational -no intervention)

SUMMARY:
Patient Registration Study of Acute Ischemic Stroke/transient ischemic attack(TIA) With Atrial Fibrillation (AISWAF) is a single-center prospective, consecutively, observational study, was conducted in patients with acute ischemic stroke/TIA with atrial fibrillation. The aim of this study was to understand the stroke mechanism, the regularity of stroke recurrence and its influencing factors, to establish a risk stratification model for stroke recurrence, and to preliminarily explore the relationship between stroke mechanism, risk stratification and antithrombotic regimen in this population.

DETAILED DESCRIPTION:
Patients with acute ischemic stroke (IS) and atrial fibrillation (AF) are at particularly high risk of recurrent IS and other major vascular events. Current antithrombotic therapy guidelines recommend oral anticoagulation (OAC) alone for the secondary prevention of IS in this high-risk population. However, these guidelines are largely based on evidence from randomized-controlled trials that did not include patients with acute IS. With the exception of the European Atrial Fibrillation Trial (EAFT), all randomized-controlled trials evaluating antithrombotic therapy in patients with AF included primary prevention populations. Moreover, the EAFT trial does not inform the management of patients with severe stroke, as these patients were excluded from this trial, and it did not evaluate the safety and efficacy of combination OAC and antiplatelet therapy.Current observational studies also provide very limited information about the optimal antithrombotic regimen for different stroke mechanisms in acute ischemic stroke/transient ischemic attack(TIA) with atrial fibrillation. In fact , the regularity of recurrence, the specific mechanism of ischemic stroke and the optimal antithrombotic regimen for different stroke mechanisms in these patients are still not clear, which limited clinical treatment level of these patients. Patient Registration Study of Acute Ischemic Stroke/transient ischemic attack(TIA) With Atrial Fibrillation (AISWAF) is a single-center prospective, consecutively, observational study, was conducted in patients with acute ischemic stroke/TIA with atrial fibrillation. The aim of this study was to understand the stroke mechanism, the regularity of stroke recurrence and its influencing factors, to establish a risk stratification model for stroke recurrence, and to preliminarily explore the relationship between stroke mechanism, risk stratification and antithrombotic regimen in this population.The clinical, imaging and laboratory information were collected at baseline. During the 1-year follow-up period, three months, six months and one year after admission, the patients were followed up by telephone or face-to-face to record the status of antithrombotic therapy, compliance, functional status, recurrence of ischemic stroke, intracranial hemorrhage, major extracranial hemorrhage as well as other vascular events and deaths.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old;
* Acute ischemic stroke or TIA within 14 days of onset (including patients with hemorrhagic transformation of infarction)
* Evidence of atrial fibrillation or newly discovered atrial fibrillation before onset (atrial fibrillation includes valvular and non-valvular, permanent, persistent or paroxysmal);
* Sign informed consent and consent to follow-up for 1 year.

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic Stroke/TIA With Atrial Fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of recurrent Ischemic stroke/TIA and symptomatic systemic embolism | one year
  recurrent ischemic stroke/TIA and symptomatic systemic embolism

SECONDARY OUTCOMES:
The rate recurrent Ischemic stroke/TIA | one year
  Recurrent ischemic stroke/TIA is defined as a new focal neurological deficit of sudden onset lasting at least 24 h (or<24 h if following therapeutic intervention, i.e. thrombolysis or thrombectomy, or if the deficit results in death< 24 h), occurring>24 h after the index ischemic stroke, irrespective of vascular territory and that is not attributable to oedema, brain shift, haemorrhagic transformation, intercurrent illness, hypoxia or drug toxicity;
The rate of symptomatic intracranial hemorrhage | one year
  Symptomatic intracranial hemorrhage(ICH) is defined as a new focal neurological deficit of sudden onset lasting at least 24 h with documented ICH on imaging (CT orMRI). Any intraparenchymal hematoma (≥ 10 mm) will be considered, including haemorrhagic transformation of the index ischemic stroke. However, microhaemorrhages (< 10 mm) do not fulfil the study definition of ICH. ICH will be classified as symptomatic if it is associated with≥4 points increase in total National Institutes of Health stroke scale (NIHSS) or≥2 points increase in 1 of the NIHSS categories ;
The rate of non-intracranial major hemorrhage | one year
  non-intracranial major hemorrhage are those that result in death or are life-threatening as defined by the International Society on Thrombosis and Haemostasis (ISTH) or consume major healthcare resources, which include: - fatal bleeding; and/or - symptomatic bleeding in a critical area or organ, such as intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome; and/or - bleeding causing a fall in haemoglobin level of≥ 20 g/L, or leading to transfusion of two or more units of whole blood or red cells; and/or - bleeding events leading to hospitalisation (in addition to the original ISTH definition)
the rate of hemorrhagic transformation and the rate of symptomatic hemorrhagic transformation | one month
  Hemorrhagic transformation (HT) was deﬁned on CT scan as any degree of hyperdensity within the area of low attenuation and was classiﬁed as either hemorrhagic infarction or parenchymal hematoma;symptomatic haemorrhagic transformation of the index ischemic stroke which is associated with≥4 points increase in total National Institutes of Health stroke scale (NIHSS) or≥2 points increase in 1 of the NIHSS categories
the rate of vascular death | one year
  vascular death is defined as the death caused by vascular events on the basis of which platelet-rich thrombi are formed
All cause death | one year
  All cause death is defined as the death from various causes
the rate of clinically relevant nonmajor bleeding | one year
  Clinically relevant nonmajor bleeding is defined as non major bleeding. resulting in hospitalization, medical or surgical intervention, or change, interruption, or discontinuation of the antithrombotic drug
Neurological disability | one year
  Neurological disability is measured with modified ranking scale (0-5). 0:No symptoms at all; 1:Despite symptoms, it has no obvious dysfunction and can perform all daily duties and activities; 2:Mild disability, unable to complete all pre-illness activities, but without help, can take care of their own affairs;3:Moderate disability requires some help, but walking does not require help; 4:Severe disability, can not walk independently, without the help of others can not meet their own needs; 5:Severe disability, bedridden, incontinence, continuous care and attention are required.
the rate of medication persistence with OAC therapy | one year
  Medication persistence with OAC therapy is defined as the absence of are fill gap of >60 days (non-persistence was defined as a gap of >60 days after the end of the day's supply of the medication of interest). Discontinuation was defined as no additional refill of the medication of interest for >90 days through to the end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sufang Xue, Beijing, Beijing Municipality, China